CLINICAL TRIAL: NCT04551495
Title: Neoadjuvant Study of Targeting ROS1 in Combination With Endocrine Therapy in Invasive Lobular Carcinoma of the Breast
Brief Title: Neoadjuvant Study of Targeting ROS1 in Combination With Endocrine Therapy in Invasive Lobular Carcinoma of the Breast (ROSALINE)
Acronym: ROSALINE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IJB-LOB-2019
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-04

CONDITIONS: Invasive Lobular Breast Carcinoma; ER+ Breast Cancer; HER2-negative Breast Cancer
MeSH Terms: conditions — Carcinoma, Lobular | interventions — entrectinib; Letrozole; Goserelin

STUDY DESIGN:
Intervention Model Description: Single arm, muti-center, phase 2 trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Subjects will receive four 28-day cycles of letrozole 2.5 mg daily in combination with entrectinib 600 mg daily. Pre-menopausal women will receive goserelin 3.6 mg every 28 days.
  Interventions: Drug: Entrectinib; Drug: Letrozole; Drug: Goserelin

INTERVENTIONS:
Drug: Entrectinib — Entrectinib is administered orally at a dose of 600 mg once a day from days 1 to 28 of a 28-day cycle for four cycles
Drug: Letrozole — Letrozole is administered orally at a dose of 2.5 mg once a day from days 1 to day 28 of a 28 day cycle for four cycles
Drug: Goserelin — Goserelin is administered subcutaneously at a dose of 3.6 mg at the beginning of each cycle for 4 monthly cycles to pre-menopausal women

SUMMARY:
Despite different clinical characteristics including the response to treatment and the patterns of metastatic relapse, invasive lobular breast carcinoma (ILBC) is treated like invasive ductal breast carcinoma (IDBC) carcinoma both in the clinics and in clinical trials. A large majority of ILBC are ER+/HER2- and almost 90% have loss of E-cadherin (CDH1) expression. A non-clinical study of CDH1 synthetic lethality interactions has identified ROS1 as a potential target. In vivo, ROS1 inhibitors produced profound antitumor effects in multiple models of E-cadherin-defective breast cancer, providing the preclinical rationale for assessing ROS1 inhibitors in this setting. Endocrine therapy being the mainstay of therapy for ER+/HER2- ILBC and the pre-operative setting offering a platform for rapid drug evaluation and biomarker research, the ROSALINE phase 2 study will evaluate the efficacy of Entrectinib (a potent inhibitor of ROS1 among other targets) in combination with letrozole (+ goserelin in premenopausal women) in the early setting of ILBC (stages 1 to 3). The neoadjuvant therapy will last 4 months and post-operative therapy will follow local practice. Biomarker research will include RNA sequencing of initial biopsies and surgical specimens, as well as liquid biopsies.

DETAILED DESCRIPTION:
The neoadjuvant setting has been the target of increasing interest recently, as it offers the possibility of direct evaluation of treatment effect on tumour size, better surgical results as well as for the possible research opportunities it provides via the comparative analysis of tumour biology and clinical outcomes before and after treatment.

Invasive lobular breast cancer (ILBC) is the second most common histologic subtype (5-15%) after invasive ductal breast cancer (IDBC). Despite clinical and pathologic differences, ILBC is still treated as IDBC. Indeed, subjects with ILBC tend to have lower response rates to conventional chemotherapeutic agents and some results have suggested that they might derive increased benefit with aromatase inhibitors.

CDK4/6 inhibitors in combination with endocrine therapy are FDA-approved for the treatment of ER-positive/HER2-negative metastatic breast cancer following the results of 7 positive phase 3 trials. These agents are currently tested in phase 3 studies in the adjuvant setting and might achieve the status of standard of care for subjects with ER-positive/HER2-negative early breast cancer treated with curative intent. In the NeoPAL (UCBG10/4, NCT02400567) neoadjuvant randomized study, Residual Cancer Burden (RCB) 0-1 status was achieved for 7.7% of subjects in the letrozole + palbociclib arm. This rate is not available for the 7 subjects with lobular breast cancer enrolled in this arm.

In lobular breast cancer, loss of E-cadherin (CDH1) expression is the most frequent oncogenic event and is present in 90% of cases. In vitro, ex vivo, and in vivo model systems as well as different functional profiling modalities (genetic and chemical screens) have been used to identify CDH1 synthetic lethality interactions. In vivo, ROS1 inhibitors produced profound antitumor effects in multiple models of E-cadherin-defective breast cancer, providing the preclinical rationale for assessing ROS1 inhibitors in this setting. A study is currently investigating this hypothesis in ER+/HER2- metastatic lobular breast cancer (NCT03620643).

Entrectinib is a potent small-molecule tyrosine kinase inhibitor that targets oncogenic rearrangements in NTRK, ROS1, and ALK. In vitro, entrectinib potently ROS1 at low nanomolar concentrations, with an average median inhibitory concentration of 0.007 μM against ROS1.

This single arm, multi-center, phase 2 trial will include pre and post-menopausal women with ER-positive/HER2-negative early stage invasive lobular carcinoma of the breast to evaluate the effect of combining endocrine therapy with entrectinib. Subjects will receive four 28-day cycles of letrozole 2.5 mg daily in combination with entrectinib 600 mg daily. Pre-menopausal women will receive goserelin 3.6 mg every 28 days.

Subjects' response to therapy will be evaluated at screening, after 2 cycles and after the 4 cycles of treatment by breast magnetic resonance imaging (MRI). An ECG will be performed at screening and then before cycle 2. Surgery will take place after at least 16 weeks of treatment, during week 18 (+ 7-day window). Breast and axillary surgery will follow local practice.

Post-operative therapy will be at the discretion of the investigator and will follow local practice.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Age ≥ 18 years
3. Histological diagnosis of invasive lobular breast adenocarcinoma that is ER+, and HER2- as per the updated American Society of Clinical Oncology (ASCO) - College of American Pathologists (CAP) guidelines according to local testing.
4. Multifocal unilateral or bilateral breast adenocarcinoma tumours are allowed if all tested foci are lobular, ER+ and HER2-.

   * ER positive (ER+ is defined as having an IHC of 1% or more and/or an Allred of 3 or more and HER2-).
   * HER2 negative as defined by 2018 ASCO / CAP Guidelines
5. A primary non metastatic or locally advanced tumour of 15 mm or more, cN0 or cN1 without prior treatment candidate for preoperative treatment.
6. ECOG Performance Status (PS) 0 or 1.
7. Adequate Bone Marrow Function including:

   * Absolute Neutrophil Count (ANC) ≥1500/μL or ≥1.5x109/L;
   * Platelets ≥100000/μL or ≥100 x 109/L;
   * Haemoglobin ≥ 9 g/dL.
8. Adequate Renal Function including:

   o Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or estimated creatinine clearance ≥ 60 ml/min as calculated using the method standard for the institution.
9. Adequate Liver Function, including all of the following parameters:

   * Total serum bilirubin ≤ 2.0 x ULN unless the subject has documented Gilbert syndrome
   * Aspartate and Alanine Aminotransferase (AST and ALT) ≤ 3 x ULN;
10. Signed Informed Consent form (ICF) obtained prior to any study related procedure.
11. Completion of all necessary screening procedures within 28 days prior to enrolment. Biopsies at screening must have been obtained up to max 6 weeks before the beginning of treatment.
12. Subject is willing and able to comply with the protocol for the duration of the study including treatment and scheduled visits and examinations.
13. Women who are not postmenopausal or have not undergone hysterectomy must have documented negative pregnancy test (serum) within 28 days prior to enrolment.
14. Women of childbearing potential and their partners, who are sexually active, must agree to use one highly effective form of contraception (see protocol section 6.6.1) from the signing of the ICF until at least 5 weeks after last administration of entrectinib, or they must totally/truly abstain from any form of sexual intercourse. Use of oral hormonal contraceptive agents in this study is not permitted.

    Inclusion criterion applicable to FRANCE only:
15. Subject is affiliated to the French Social Security System.

Exclusion Criteria:

1. Clinical T4 disease including inflammatory breast cancer and/or cN3.
2. Prior history of invasive cancer in the past 5 years except basal or squamous cell carcinoma of skin that has been definitively treated.
3. Known hypersensitivity to the study drugs or excipients.
4. Hyperuricemia > Grade 1
5. Any illness or medical condition that is unstable or could jeopardize the safety of the subject or her compliance with study requirements.
6. Subjects unable to swallow oral medications.
7. Prior intake of letrozole, any ROS1 inhibitor, any TRK inhibitor or anticancer therapy (including endocrine therapy). Ovarian suppression including prior administration of a LHRH analogue (i.e. goserelin) is allowed prior to cycle 1 day 1, at the discretion of the investigator.
8. Concurrent treatment with strong or moderate CYP3A inhibitor.
9. Concurrent treatment with any of the drugs not permitted, i.e. strong CYP3A inducers and drugs known to cause QTc interval prolongation.
10. Significant cardiac disease, including recent (less than 6 months) myocardial infarction, congestive heart failure, unstable angina, and bradyarrhythmias.
11. LVEF ≤ 55% measured by echo or MUGA
12. QTc exceeding 450 msec, history of prolonged QTc interval prolongation; risk factors for torsade de pointes; other concomitant medications that may prolong QTc; family or personal history of long or short QT syndrome, Brugada syndrome or known history of QTc prolongation, or Torsade de Pointes (TdP).
13. Pregnant or lactating women.
14. Known interstitial lung disease, interstitial fibrosis, or history of tyrosine kinase inhibitor-induced pneumonitis
15. Peripheral neuropathy ≥ Grade 2
16. Active gastrointestinal disease (e.g., Crohn's disease, ulcerative colitis, or short gut syndrome) or other malabsorption syndromes that would reasonably impact drug absorption.

    Exclusion criterion applicable to France only
17. Vulnerable persons according to the article L.1121-6 of the CSP, adults who are the subject of a measure of legal protection or unable to express their consent according to article L.1121-8 of the CSP.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 65 (Estimated)
Dates: Start 2021-01-14 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the efficacy of endocrine therapy + entrectinib in women with ER+/HER2- early breast cancer of the lobular subtype:Residual Cancer Burden (RCB) | At surgery
  Residual Cancer Burden (RCB) 0/1 by local evaluation in all enrolled subjects.

SECONDARY OUTCOMES:
Evaluation of the efficacy of the combination by pathology: Pathologic complete response (pCR) rate | At surgery
  Pathologic complete response (pCR) rate in breast and axilla (ypT0/Tis ypN0) by local evaluation

OTHER OUTCOMES:
Evaluation the efficacy of the combination by imaging: Tumour objective response | At surgery
  Tumour objective response assessed by locally-assessed breast MRI via modified Response Evaluation Criteria in Solid Tumours (RECIST 1.1.)
Evaluation of the safety of endocrine therapy + entrectinib: adverse events | Up to 5 months
  Incidence, nature, and severity of adverse events graded according to National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (NCI CTCAE, v5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Aftimos, MD, Study Chair — Jules Bordet Insitute
Locations (10):
- Belgium (7):
  - Institut Jules Bordet, Brussels
  - UZ Brussel, Brussels
  - UCL Saint-Luc, Brussels
  - Grand Hôpital de Charleroi, Charleroi
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - CHU Namur - Sainte Elisabeth, Namur
- France (3):
  - Institut Bergonié, Bordeaux
  - Institut Curie, Paris
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Agostinetto E, Nader-Marta G, Paesmans M, Ameye L, Veys I, Buisseret L, Neven P, Taylor D, Fontaine C, Duhoux FP, Canon JL, Denys H, Coussy F, Chakiba C, Ribeiro JM, Piccart M, Desmedt C, Ignatiadis M, Aftimos P. ROSALINE: a phase II, neoadjuvant study targeting ROS1 in combination with endocrine therapy in invasive lobular carcinoma of the breast. Future Oncol. 2022 Jul;18(22):2383-2392. doi: 10.2217/fon-2022-0358. Epub 2022 Jun 13. PMID 35695563
- [Derived] Okines A, Irfan T, Asare B, Mohammed K, Osin P, Nerurkar A, Smith IE, Parton M, Ring A, Johnston S, Turner NC. Clinical outcomes in patients with triple negative or HER2 positive lobular breast cancer: a single institution experience. Breast Cancer Res Treat. 2022 Apr;192(3):563-571. doi: 10.1007/s10549-021-06432-z. Epub 2022 Feb 4. PMID 35119530